CLINICAL TRIAL: NCT06864676
Title: Assessment of the Diagnostic Performance of the Detection System and Establishment of an Intelligent and Rapid Triage Model
Status: Not yet recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023YFC2413005; 2023YFC2413005 (Other: Ministry of Science and Technology of the People's Republic of China)
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Coronary Heart Disease (CHD)
Keywords: ACS
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Plasma or serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The rapid triage of patients with acute chest pain remains an important issue in clinical practice. This study will establish a cohort of patients suspected of acute coronary syndrome (ACS) to construct a multi-marker dynamic combined intelligent triage model. This model will triage the risk of NSTEMI in patients with chest pain at their first visit. It will also stratify the risk of patients with chest pain using major adverse cardiovascular events (MACE) within 30 days as the endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or above from China, regardless of gender;
* Presence of symptoms such as chest tightness and chest pain, with the need to determine whether they are patients with acute coronary syndrome;
* Ability to obtain informed consent.

Exclusion Criteria:

* - Patients with STEMI at the time of presentation;
* Patients with a clear diagnosis after tests such as troponin;
* Patients who have undergone major surgery or trauma within the past four weeks;
* Pregnant women or patients with tumors undergoing radiotherapy or chemotherapy;
* Patients who have previously participated in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese population aged 18 years and above, regardless of gender, with symptoms of chest tightness and chest pain, who need to be confirmed as acute coronary syndrome patients.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Myocardial infarction | 30 days to 6 months
  in patients suspected of NSTEMI, using the baseline (0 hours) and any one of the 1-3 hour points for the ZR iStar (POCT) hs-cTnI two-point method, combined with the time from typical chest pain to the visit, to establish a triage machine learning model for NSTEMI through the training cohort, and to establish a multi-marker dynamic combination intelligent triage model for risk stratification of chest pain patients.

OTHER OUTCOMES:
High-sensitivity troponin | Concentrated detection once every three months
  Validation of instruments and test kits by detecting high-sensitivity troponin levels using different platforms.